CLINICAL TRIAL: NCT00326053
Title: A Comparison of Budesonide/Formoterol Turbuhaler® 160/4.5 µg 2 Inhalations BID Plus as Needed to Budesonide Turbuhaler® 320 µg 2 Inhalations BID Plus Terbutaline Turbuhaler® 0.4 mg as Needed for the Prevention of Asthma Relapse
Brief Title: Prevention of Asthma Relapse After Discharge From Emergency
Acronym: PARADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5890L00017; PARADE
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma Reoccurrence; Acute Asthma; Patient Discharge; Emergency Service, Hospital; Asthma Exacerbation; Asthma Relapse
MeSH Terms: conditions — Asthma; Emergencies | interventions — Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol
  Other Names: Symbicort

SUMMARY:
The purpose of this study is to compare the Symbicort® Turbuhaler® to both Pulmicort® Turbuhaler® and Bricanyl® Turbuhaler® for the treatment of asthma after discharge from the emergency room

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age
* Presenting at a study emergency department with an asthma exacerbation

Exclusion Criteria:

* Admission to hospital
* Patients receiving more than 2000 µg/day of beclomethasone equivalent inhaled corticosteroids (1000 µg/day fluticasone or 1600 µg/day budesonide)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Time to first asthma relapse

SECONDARY OUTCOMES:
Mean use of reliever medication
Asthma Control Questionnaire (ACQ) score
Complete AE and SAE collection

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Jordana, MD, Study Director — AstraZeneca; Brian Rowe, MD, Principal Investigator — University of Alberta
Locations (20):
- Canada (20):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Lethbridge, Alberta
  - Research Site, St. Albert, Alberta
  - Research Site, Nanaimo, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Truro, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, La Malbaie, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Ste-Foy, Quebec
  - Research Site, Saskatoon, Saskatchewan